



Mr Daniel Howgate

Honorary Specialty Registrar Trauma & Orthopaedic Surgery and DPhil Student Botnar Institute of Musculoskeletal Sciences, University of Oxford, Old Road, Oxford, OX3 7LD

E-mail: daniel.howgate@ndorms.ox.ac.uk Oxford telephone number: 01865 760063

| | SURGEON PARTICIPANT CONSE | ENT FORM: SPECIALTY REGISTRA | RS |
|---|---|---|---|
| lρ | | y assessing surgical performance and the aining in primary THR | impact |
| | · | anning in primary raik | |
| Var | ne of Researcher: | If you agree, please initial | box |
| 1. | I confirm that I have read the information | sheet dated (version) | |
| | for this study. I have had the opportunity to consider the information, ask questions | | |
| | and have had these answered satisfactorily. | | |
| <b>1</b> | | stani, and that I am for a to with discuss to an | |
| 2. | time without giving any reason. | ntary and that I am free to withdraw at any | |
| | time without giving any reason. | | |
| 3. | I understand that relevant sections of my anonymised data collected during the | | |
| | study may be looked at by individuals from University of Oxford, from regulatory | | |
| | authorities and from the NHS Trust(s), where it is relevant to my taking part in this | | |
| | research. I give permission for these individuals to have access to my records. | | |
| 4. | I understand that responsible members of the research team may request sections of | | |
| | my training data (e.g. 'logbook' or ePortfolio) and link this to my anonymized | | |
| | research data where it is relevant to my taking part in this research. I give permission | | |
| | for these individuals to use such data I provide. | | |
| | I agree to take part in this study. | | |
| 5. | | | |

Surgeon Participant Consent form: StR THR Performance & Assessment Professor Jonathan Rees

Version 2.0 12th October 2019 IRAS Project number: 270167 REC Reference number: 19/SC/0492

| Name of Person | taking |
|----------------|--------|
| Consent | |

Date

Signature

\*1 copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes (if participant is a patient).

Surgeon Participant Consent form: StR THR Performance & Assessment Professor Jonathan Rees Version 2.0 12<sup>th</sup> October 2019 IRAS Project number: 270167 REC Reference number: 19/SC/0492